CLINICAL TRIAL: NCT01076465
Title: Efficacy of a Disease Management Program in Very Old Patients With Heart Failure and Significant Comorbidity: a Multicenter Randomized Trial
Brief Title: Efficacy of a Disease Management Program in Very Old Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Meixoeiro (Other Government)
Collaborators: Complejo Hospitalario Universitario de Vigo (Other); Universidad Autonoma de Madrid (Other); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Carlos RodrÃ-guez Pascual, MD, PhD, Hospital de Meixoeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI081280; PI081280 (Other Grant/Funding Number: Fondo de Investigación Sanitaria, Spain)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure; Comorbidity; Case-manager
Keywords: Heart failure; Elderly; Disease management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counselling (Experimental): Educational intervention, monitoring of clinical status, monitoring of treatment adherence
  Interventions: Other: Disease management program
- Comparator (Active Comparator): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Other: Disease management program — 1. Educational intervention on management of heart failure and comorbidity to improve patient's knowledge of his/her disease and self-care 2) Monitoring of clinical status 3) Monitoring and improvement of therapeutic adherence.
  Arms: Lifestyle counselling
Behavioral: Usual care — Usual care
  Arms: Comparator

SUMMARY:
The purpose of this study is to assess the efficacy of a disease management programme (DMP) for very old patients with HF and significant co-morbidity.

METHODS: A multicenter randomized trial will be conducted with 700 patients with heart failure, aged over 75 years, admitted to the acute-care units of the Geriatrics Departments in 8 hospitals. Patients will be randomly allocated to a DMP or to conventional usual-care. Randomization will be stratified by hospital and performed with concealment of the allocation list.

The DMP will be conducted by a case manager, and will include three main components:

1. patient education to improve disease' knowledge and self-care
2. monitoring of clinical status
3. therapeutic adherence. Main statistical analyses will be performed according to the intention-to-treat principle, and will use Cox regression models to examine the association of a DMP with hospital readmission, quality-of-life, and mortality over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age:75 y or older
2. Co-morbidity or dependency. At least one of the following criteria: Charlson index >3, dependency in 2 or more basic activities of daily living,treatment with 5 or more drugs, urgent hospitalization in the last 3 months, three or more diseases with active treatment, limitation in daily living because of vision or hearing impairment, cognition deficit, Parkinson disease, diabetes mellitus, chronic obstructive lung disease, severe anemia, constitutional syndrome
3. Hospital admission with a main diagnosis of heart failure (according to the criteria of the European Society of Cardiology or Framingham criteria) in NYHA functional class II-IV.

Exclusion Criteria:

1. Participation refusal
2. Terminal illness
3. Cognitive decline or severe cognitive deficit, which does not permit a minimum knowledge of the disease, or lack of carers which give consent to study participation
4. Clinical instability as assessed with the Kosecof index
5. Being in waiting list for organ transplant or cardiac surgery
6. Inability to be followed-up because of other reasons (change of place of residence,..)
7. Institutionalization

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 700 (Actual)
Dates: Start 2009-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mortality or readmission | one year

SECONDARY OUTCOMES:
Health related quality of life | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Meixoeiro, Vigo, Pontevedra, Spain

REFERENCES:
- [Derived] Pascual CR, Galan EP, Guerrero JL, Colino RM, Soler PA, Calvo MH, Jaurieta JJ, Arambarri JM, Casado JM, Rodriguez-Artalejo F. Rationale and methods of the multicenter randomised trial of a heart failure management programme among geriatric patients (HF-Geriatrics). BMC Public Health. 2011 Aug 5;11:627. doi: 10.1186/1471-2458-11-627. PMID 21819564